CLINICAL TRIAL: NCT04593914
Title: Evaluating the Effectiveness of a Novel Skin Barrier Protectant in the Prevention and Management of Acute Radiodermatitis in Patients With Head and Neck Cancer: a Prospective Cohort Study With Historical Controls
Brief Title: A Novel Skin Barrier Protectant for Acute Radiodermatitis
Acronym: CASP-ORL
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid-19
Sponsor: Jessa Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20.17-ONCO20.04
Record Dates: First submitted 2020-10-08; First posted 2020-10-20 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Radiodermatitis; Radiation Toxicity; Radiation Dermatitis; Skin Diseases; Head and Neck Cancer
MeSH Terms: conditions — Radiodermatitis; Radiation Injuries; Skin Diseases; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cavilon Advanced Skin Protectant (Experimental): Cavilon Advanced Skin Protectant forms a film barrier intended to protect intact or damaged skin. It is effective in conditions where skin is frequently or continuously exposed to moisture and caustic irritants such as feces, digestive fluids, wound drainage and urine. Cavilon Advanced Skin Protectant also can be used in areas exposed to friction and shear from bedding, clothing, shoes or any other material that would rub against the skin.
  The skin barrier protectant will be applied on the irradiated skin from the third week of radiotherapy until 1 week after the final radiotherapy session.
  Interventions: Device: Cavilon Advanced Skin Protectant

INTERVENTIONS:
Device: Cavilon Advanced Skin Protectant — 3M™ Cavilon™ Advanced Skin Protectant is a polymeric-cyanoacrylate solution intended for the protection of intact or damaged skin. Upon application to skin, the liquid dries rapidly to form a primary long-lasting waterproof, highly durable film barrier. It is elastomeric, adhering to the contours of the skin and providing a uniform film. The film is transparent and possesses good oxygen and moisture vapor permeability.
  The polymer-cyanoacrylate is dispersed in a non-stinging solvent. The film is colorless, non-cytotoxic and has a low dermatitis potential. The film adheres to dry, moist or wet skin surfaces and remains intact during conditions of continuous or repeated exposure to moisture or caustic irritants. It will wear off the skin and does not require removal.

SUMMARY:
Acute radiodermatitis (ARD) is a distressing and painful skin reaction that occurs in 95% of the patients undergoing radiotherapy (RT). To date, there is still no general approved guideline for the prevention and management of acute radiodermatitis. The 3M™ Cavilon™ Advanced Skin Protectant is a novel skin barrier protectant that acts as a physical barrier against abrasion, moisture, and irritants. Moreover, it enables an environment for wound healing. The aim of this study is to evaluate the effectiveness of 3M™ Cavilon™ Advanced Skin Protectant in the prevention and management of ARD in patients with head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of head and neck squamous cell carcinomas (HNSCC) starting in the lip, salivary gland, oral cavity (mouth), nasal cavity (inside the nose), paranasal sinuses, pharynx, or larynx.
* Scheduled for bilateral neck radiotherapy (>60 Gy) with or without concomitant chemotherapy either as primary or as post-operative treatment to the head and neck region
* Age ≥ 18 years
* Able to comply to the study protocol
* Able to sign written informed consent
* Signed written informed consent

Exclusion Criteria:

* Previous irradiation to the head and/or neck region
* Metastatic disease
* Patients with pre-existing skin rash, ulceration or open wound in the treatment area
* Patients with known allergic and other systemic skin diseases even when not directly affecting irradiated fields
* Substance abuse patients or patients with medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results as judged by the investigator
* Any condition that is unstable or could affect the safety of the patient and their compliance in the study as judged by the investigator
* Patients using high doses of non-steroidal anti-inflammatory drugs
* Patients allergic to the ingredients of the 3M™ Cavilon™ Advanced Skin Protectant

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Radiodermatitis grading | Day 1
  National Cancer Institute-Common Terminology Criteria for Adverse Events version 4.03
Radiodermatitis grading | Day 14
  National Cancer Institute-Common Terminology Criteria for Adverse Events version 4.03
Radiodermatitis grading | Day 20
  National Cancer Institute-Common Terminology Criteria for Adverse Events version 4.03
Radiodermatitis grading | Day 35
  National Cancer Institute-Common Terminology Criteria for Adverse Events version 4.03
Radiodermatitis grading | Day 38
  National Cancer Institute-Common Terminology Criteria for Adverse Events version 4.03
Radiodermatitis grading | Day 47
  National Cancer Institute-Common Terminology Criteria for Adverse Events version 4.03
Radiodermatitis severity | Day 1
  Radiation-Induced Skin Reaction Assessment Scale (0- 36, with a higher score correlating with a more severe skin reaction)
Radiodermatitis severity | Day 14
  Radiation-Induced Skin Reaction Assessment Scale (0- 36, with a higher score correlating with a more severe skin reaction)
Radiodermatitis severity | Day 20
  Radiation-Induced Skin Reaction Assessment Scale (0- 36, with a higher score correlating with a more severe skin reaction)
Radiodermatitis severity | Day 35
  Radiation-Induced Skin Reaction Assessment Scale (0- 36, with a higher score correlating with a more severe skin reaction)
Radiodermatitis severity | Day 38
  Radiation-Induced Skin Reaction Assessment Scale (0- 36, with a higher score correlating with a more severe skin reaction)
Radiodermatitis severity | Day 47
  Radiation-Induced Skin Reaction Assessment Scale (0- 36, with a higher score correlating with a more severe skin reaction)

SECONDARY OUTCOMES:
Quality of life measurement | day 1
  Patient's quality of life will be assessed by using Skindex-16
Quality of life measurement | day 14
  Patient's quality of life will be assessed by using Skindex-16
Quality of life measurement | day 20
  Patient's quality of life will be assessed by using Skindex-16
Quality of life measurement | day 35
  Patient's quality of life will be assessed by using Skindex-16
Quality of life measurement | day 38
  Patient's quality of life will be assessed by using Skindex-16
Quality of life measurement | day 47
  Patient's quality of life will be assessed by using Skindex-16
General satisfaction | Day 35
  Patients' general satisfaction with the skin barrier will be evaluated by using a self-developed questionnaire
General satisfaction | day 38
  Patients' general satisfaction with the skin barrier will be evaluated by using a self-developed questionnaire
General satisfaction | day 47
  Patients' general satisfaction with the skin barrier will be evaluated by using a self-developed questionnaire

OTHER OUTCOMES:
Clinical photograph | day 1
  A clinical photograph of the treatment area will be taken
Clinical photograph | day 14
  A clinical photograph of the treatment area will be taken
Clinical photograph | day 20
  A clinical photograph of the treatment area will be taken
Clinical photograph | day 35
  A clinical photograph of the treatment area will be taken
Clinical photograph | day 38
  A clinical photograph of the treatment area will be taken
Clinical photograph | day 47
  A clinical photograph of the treatment area will be taken
Personal and medical information | day 1
  Patient's personal and medical information will be gathered via a patient questionnaire and the patient's medical file

CONTACTS AND LOCATIONS:
Overall Officials: Annelies Maes, MD, Principal Investigator — Limburgs Oncologisch Centrum
Locations (2):
- Belgium (2):
  - Ziekenhuis Oost-Limburg, Genk, Limburg
  - Jessa Ziekenhuis, Hasselt, Limburg

IPD SHARING:
Plan to Share IPD: No